CLINICAL TRIAL: NCT03213535
Title: Urea and Creatinine Level in Vaginal Fluid as a Predicator for Length of Latency Period in Prelabour Membranes Rupture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, rasha medhat abdul-hady, principal Investigator Dr.rasha medhat abdul-hady, Ain Shams University
Other Study IDs: PRP-PROM
Record Dates: First submitted 2017-07-08; First posted 2017-07-11 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-01

CONDITIONS: Rupture of Membranes; Premature
Keywords: PROM
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the relation between the concentration of urea and creatinine in vaginal fluid and length of latency period in women with PROM between 32 and 35 weeks gestation.

DETAILED DESCRIPTION:
60 pregnant women with PROM with singleton pregnancies with a gestational age between 32- 35 gestational weeks History taking followed by examination All women will be put in dorsal lithotomy position, using a proper light source and sterile gloves; sterile speculum free of gel will be placed into vagina.

For every woman a specimen of vaginal fluid will be taken as follows: 5 ml of sterile saline solution will be injected into the posterior vaginal fornix taken after aspiration of 3ml with the same syringe.

All samples will be obtained within 6 hours after membranes rupture before vaginal examination and the administration of any drugs. Upon collection, samples were centrifuged at 3000 rpm for 10 minutes and supernatant fluid was separated. Exact concentrations of urea and creatinine will be measured

All women will be put under observation for 48 hours and time of onset of delivery will be documented, the onset of labor will be diagnosed by either:

1. Frequent uterine contractions more than 2 contractions in 10 minutes.
2. CTG showing frequent contractions.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age between 20-35 years.
2. 32-35 weeks gestational age.
3. Viable fetus.

Exclusion Criteria:

1. Vaginal bleeding either spontaneous or traumatic e.g. placenta previa.
2. Chorioamnionitis.
3. Multiple pregnancy.
4. Presence of uterine contractions.
5. Amniotic fluid disorders e.g. polyhydramnios
6. Meconium stained amniotic fluid prior to active phase of labor.
7. Maternal disease necessitating termination of pregnancy e.g. severe preeclampsia

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: sixity pregnant women with PROM with singleton pregnancies with a gestational age between 32- 35 gestational weeks by reliable menstrual history and confirmed by pelvi-abdominal ultrasound.
  Membranes rupture will be diagnosed by the direct visualization of fluid leakage from the cervical canal using sterile speculum.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-07-10 (Estimated); Study Completion 2017-07-10 (Estimated)

PRIMARY OUTCOMES:
delivery interval in Premature rupture of membranes | 48 hours
  The time needed from the onset of PROM till time of onset of labour

CONTACTS AND LOCATIONS:
Overall Officials: rasha M Medhat Abd El-Hady, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dare MR, Middleton P, Crowther CA, Flenady VJ, Varatharaju B. Planned early birth versus expectant management (waiting) for prelabour rupture of membranes at term (37 weeks or more). Cochrane Database Syst Rev. 2006 Jan 25;(1):CD005302. doi: 10.1002/14651858.CD005302.pub2. PMID 16437525
- [Background] Gezer C, Ekin A, Golbasi C, Kocahakimoglu C, Bozkurt U, Dogan A, Solmaz U, Golbasi H, Taner CE. Use of urea and creatinine levels in vaginal fluid for the diagnosis of preterm premature rupture of membranes and delivery interval after membrane rupture. J Matern Fetal Neonatal Med. 2017 Apr;30(7):772-778. doi: 10.1080/14767058.2016.1188072. Epub 2016 May 26. PMID 27160546
- [Background] Kafali H, Oksuzler C. Vaginal fluid urea and creatinine in diagnosis of premature rupture of membranes. Arch Gynecol Obstet. 2007 Mar;275(3):157-60. doi: 10.1007/s00404-006-0240-1. Epub 2006 Sep 12. PMID 16967274
- [Background] Kim YH, Park YW, Kwon HS, Kwon JY, Kim BJ. Vaginal fluid beta-human chorionic gonadotropin level in the diagnosis of premature rupture of membranes. Acta Obstet Gynecol Scand. 2005 Aug;84(8):802-5. doi: 10.1111/j.0001-6349.2005.00712.x. PMID 16026409
- [Background] Melamed N, Hadar E, Ben-Haroush A, Kaplan B, Yogev Y. Factors affecting the duration of the latency period in preterm premature rupture of membranes. J Matern Fetal Neonatal Med. 2009 Nov;22(11):1051-6. doi: 10.3109/14767050903019650. PMID 19900043
- [Background] Ngwenya S, Lindow SW. 24 hour rhythm in the timing of pre-labour spontaneous rupture of membranes at term. Eur J Obstet Gynecol Reprod Biol. 2004 Feb 10;112(2):151-3. doi: 10.1016/s0301-2115(03)00286-0. PMID 14746949
- [Background] Oliveira FR, Barros EG, Magalhaes JA. Biochemical profile of amniotic fluid for the assessment of fetal and renal development. Braz J Med Biol Res. 2002 Feb;35(2):215-22. doi: 10.1590/s0100-879x2002000200010. PMID 11847525
- [Background] Ramsey PS, Lieman JM, Brumfield CG, Carlo W. Chorioamnionitis increases neonatal morbidity in pregnancies complicated by preterm premature rupture of membranes. Am J Obstet Gynecol. 2005 Apr;192(4):1162-6. doi: 10.1016/j.ajog.2004.11.035. PMID 15846196
- [Background] Pintucci A, Meregalli V, Colombo P, Fiorilli A. Premature rupture of membranes at term in low risk women: how long should we wait in the "latent phase"? J Perinat Med. 2014 Mar;42(2):189-96. doi: 10.1515/jpm-2013-0017. PMID 24259235
- [Background] Ramsey PS, Nuthalapaty FS, Lu G, Ramin S, Nuthalapaty ES, Ramin KD. Contemporary management of preterm premature rupture of membranes (PPROM): a survey of maternal-fetal medicine providers. Am J Obstet Gynecol. 2004 Oct;191(4):1497-502. doi: 10.1016/j.ajog.2004.08.005. PMID 15507990
- [Background] Tigga M.P. and Malik S. Comparative analysis of four biomarkers in diagnosing premature rupture of membranes and their correlation with onset of labour: Int J Reprod Contracept Obstet Gynecol. 2015 Aug;4(4):1070-1075
- [Background] Tyden O, Eriksson U, Agren H, Berne C. Estimation of fetal maturity by amniotic fluid cytology, creatinine, lecithin/sphingomyelin ratio and phosphatidylglycerol. Gynecol Obstet Invest. 1983;16(6):317-26. doi: 10.1159/000299289. PMID 6654186
- [Background] van der Ham DP, Vijgen SM, Nijhuis JG, van Beek JJ, Opmeer BC, Mulder AL, Moonen R, Groenewout M, van Pampus MG, Mantel GD, Bloemenkamp KW, van Wijngaarden WJ, Sikkema M, Haak MC, Pernet PJ, Porath M, Molkenboer JF, Kuppens S, Kwee A, Kars ME, Woiski M, Weinans MJ, Wildschut HI, Akerboom BM, Mol BW, Willekes C; PPROMEXIL trial group. Induction of labor versus expectant management in women with preterm prelabor rupture of membranes between 34 and 37 weeks: a randomized controlled trial. PLoS Med. 2012;9(4):e1001208. doi: 10.1371/journal.pmed.1001208. Epub 2012 Apr 24. PMID 22545024
- [Background] Zuo Y, Wang C, Zhou J, Sachdeva A, Ruelos VC. Simultaneous determination of creatinine and uric acid in human urine by high-performance liquid chromatography. Anal Sci. 2008 Dec;24(12):1589-92. doi: 10.2116/analsci.24.1589. PMID 19075469